CLINICAL TRIAL: NCT04704115
Title: Evaluate the Therapy of Large Ovarian Endometrioma
Brief Title: The Therapy of Large Endometrioma
Acronym: ENDOKYSTE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_43; 2020-A02354-35 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endometrioma; Endometriosis Ovary
Keywords: Endometriomas measuring 6 cm or more; Ovarian Endometrioma; laparoscopic drainage; recurrence; AMH; GnRH agonist therapy
MeSH Terms: conditions — Endometriosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrioma's prevalence is between 23 and 55%. It causes pelvic pain, decrease fertility and ovarian reserve.

Currently, there's no recommendation about large endometrioma's treatment and there's no information on the best treatment to limit recurrences, preserve fertility and ovarian reserve.

In Lille university hospital, simple laparoscopic drainage associated with hormonal therapy is practiced to reduce the risk of cystectomy.

This protocol will be evaluated with an observational and prospective study, including women of childbearing age having endometrioma measuring 6 cm or above.

The aim of this study is to assess if cyst drainage associated with GnRH agonist, could decrease endometrioma recurrences, deleterious effect on ovarian reserve and evaluate impact on anti-mullerian hormone

ELIGIBILITY:
Inclusion Criteria:

* Endometrioma size ≥ 6cm determined by MRI or ultrasonography
* Women with isolated endometrioma or other extraovarian endometriosis: peritoneal, infiltrating endometriotic lesions and adenomyosis.
* Cyst single or bilateral

Exclusion Criteria:

* Cyst with radiographic or macroscopic in laparoscopy atypia
* Pregnancy
* Patient with contraindication to GnRH agonist (Enantone® 3,75 mg et Decapeptyl® 3 mg)
* Patient with contraindication to laparoscopy
* Patient with contraindication to general anesthesia
* Subject refusing to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Study Population: Women presenting at a surgical consultation for the management of an endometrioma of 6cm or more
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Recurrence of cyst ≥ 3 cm determined by MRI or pelvic ultrasonography (US) | at 3 months

SECONDARY OUTCOMES:
The impact of the ovarian reserve postoperative | at 3 months
  Compare the dosages of anti-mullerian hormone (AMH) preoperative and postoperative at 3 months
The number of re-operation | at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Chrytèle RUBOD, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lisle-sur-Tarn, France